CLINICAL TRIAL: NCT06127095
Title: New perSEPtion. New Patient's Perspectives Beyond Clinical Efficacy of Monoclonal Antibody-Based RRMS Treatments.
Brief Title: A Study to Assess New Participant's Perspectives Beyond Clinical Efficacy of Monoclonal Antibody-Based Relapsing Remitting Multiple Sclerosis (RRMS) Treatments
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: FR-TYS-12186; 2023-A01349-36 (Other: CPP Nord Ouest)
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with RRMS: Participants who receive natalizumab intravenously (IV) or subcutaneously (SC) or ocrelizumab, or ofatumumab, as per the standard local prescribing procedures will be enrolled to collect data. Participants will complete an online one-shot questionnaire combining closed and open-ended questions.

SUMMARY:
The primary objective of the study is to understand what the added value of natalizumab (Tysabri®) treatment is from a participant's perspective at a given time, based on a one-shot survey. The secondary objectives of the study also aim to characterize the participant's decision-making process to get the treatment; the burden of treatment, characterization of the study population, assessment of the quality of life (QoL), and fatigue dimension.

ELIGIBILITY:
Inclusion Criteria:

• Participants diagnosed with RRMS and followed by a neurologist in France.

Exclusion Criteria:

• Lack of literacy

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with RRMS who have been prescribed natalizumab (Tysabri®) whether injected IV or SC, ocrelizumab (Ocrevus®), or ofatumumab (Kesimpta®) under standard clinical care for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Perceived the Treatment Added Value of Natalizumab Assessed by Likert's Scale | Day 1
  A Likert scale is a rating scale used to measure opinions, attitudes, or behaviors. This 7-pointer scale consists of a statement or a question, followed by a series of five or seven answer statements. Respondents choose the option that best corresponds with how they feel about the statement or question. The options include: strongly agree, agree, somewhat agree, neutral, somewhat disagree, disagree to strongly disagree.

SECONDARY OUTCOMES:
Number of Participants who Perceived Burden of Treatment Assessed by Closed and Open-ended Questions | Day 1
Number of Participants With Perceived Decision-making Process Assessed by Likert's Scale | Day 1
  A Likert scale is a rating scale used to measure opinions, attitudes, or behaviors. This 7-pointer scale consists of a statement or a question, followed by a series of five or seven answer statements. Respondents choose the option that best corresponds with how they feel about the statement or question. The options include: strongly agree, agree, somewhat agree, neutral, somewhat disagree, disagree to strongly disagree.
Number of Participants With Perceived Decision-making Process Assessed by Open-ended Questions on Quality of Life (QOL) | Day 1
Number of Participants Characterized by Multiple Sclerosis (MS) Types | Day 1
Number of Participants Characterized by MS Duration | Day 1
Number of Participants Characterized by Current Disease Modifying Treatment (DMT) | Day 1
Mean Multiple Sclerosis International Quality of Life Questionnaire (MusiQol) Score | Day 1
  The MusiQoL is a self-administered questionnaire consisting of 31 items describing nine dimensions of health-related QoL: activities of daily living, psychological wellbeing, symptoms, relationship with friends, relationship with family, sentimental and sexual life, coping rejection, relationship with healthcare system. All items are scored based on frequency/extent of an event on a five-point scale ranging from 1 (never/not at all) to 5 (always/very much). Total score is obtained by linearly transforming and standardizing on a 0-100 scale. Higher scores indicate a better QOL.
Mean Fatigue Severity Scale (FSS) Score | Day 1
  FSS is designed to differentiate fatigue from clinical depression. FSS is a 9-item questionnaire that requires the participant to rate their own level of fatigue on a scale of 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 9 to 63. A higher total score indicates greater fatigue severity and impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Biogen, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/